CLINICAL TRIAL: NCT02315053
Title: Dynamic FDG-PET/CT Response During Chemoradiation for NSCLC
Brief Title: PET Response During Chemoradiation of Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N12LPR
Record Dates: First submitted 2014-06-05; First posted 2014-12-11 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: NSCLC
Keywords: NSCLC; CCRT; FDG PET/CT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low dose FDG PET/CT 5x (Other): Stage II/III NSCLC will undergo a Low dose FDG PET/CT 5x during treatment (CCRT).
  Interventions: Other: Low dose FDG PET/CT 5 x.

INTERVENTIONS:
Other: Low dose FDG PET/CT 5 x. — Multiple FDG PET/CT studies will be added to the normal diagnostic procedures as a part of this study, with the number of scans depending on the study stage, to a maximum of 6 per patient.
  Other Names: No treatment intervention but diagnostic intervention.

SUMMARY:
A prospective observational study to determine the prognostic value of the timing of 50% reduction in metabolic activity (T50) during CCRT for NSCLC for treatment outcome (PFS).

DETAILED DESCRIPTION:
This is a single-centre observational study. Patients with proven locally advanced NSCLC will be treated with concurrent chemoradiotherapy according to the standard clinical protocol of the NKI-AVL. During treatment, the biological behaviour of the tumour will be monitored with serial quantitative FDG (fluorodeoxyglucose) PET/CT scans. From these images, the time during treatment where a 50% reduction in FDG uptake relative to day 1 is reached (T50) will be derived. The T50 of progression-free surviving patients will be compared with that of relapsed or deceased patients, in order to find a value that predicts early treatment failure. An additional FDG PET/CT scan at the same day as regular follow up CT scan will be made, two months after treatment, to have a baseline after treatment for follow up.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically proven NSCLC
* T2-4 N0-3 M0 disease (stage II or III, inoperable)
* Scheduled for standard concurrent chemoradiation
* Primary tumour minimal diameter 3 cm
* Primary tumour SUVmax > 5 on routine diagnostic pre-treatment FDG (Fludeoxyglucose) PET/CT
* WHO performance 0-1
* Written informed consent according to GCP (Good Clinical Practice) and national regulations

Exclusion Criteria:

* Age < 18 years, incapacitated subjects
* Pregnant or lactating women
* Diabetes mellitus requiring medication
* Participation in dose escalation studies
* Other neoplasms in the last 3 years, with metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03-21 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
maximum FDG uptake (SUVmax) | 1 Year
  • A main study parameter is the maximum FDG uptake (SUVmax (maximum Standardized Uptake Value)) at the location of the primary tumour, as determined at multiple days during treatment (with a maximum of five time points per patient), expressed as T50 for response evaluation.

SECONDARY OUTCOMES:
SUVmax during the first two weeks of treatment, indicating inflammatory response. | First Two weeks of treatment
  • Increase SUVmax during the first two weeks of treatment, indicating inflammatory response.
SUVmax in the two weeks prior to treatment, indicating progression | Two weeks prior to treatment
  • Increase SUVmax between diagnostic imaging and start of treatment, indicating potential progression.
Progression free survival | 1 Year
  • Secondary study endpoint is progression free survival, to be associated with T50 for prognostic value.

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Vogel, MD,PhD, Principal Investigator — NKI
Locations (1):
- The Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands